CLINICAL TRIAL: NCT01082783
Title: Autoimmune Phenomena After Acute Stroke - the Role of Stroke-induced Immunodepression
Brief Title: Autoimmune Phenomena After Acute Stroke
Acronym: ARIMIS
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, Andreas Meisel, Professor Dr. med., Charite University, Berlin, Germany
Other Study IDs: ARIMIS
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Stroke
Keywords: stroke-induced immunodepression; acute media infarct; acute intracerebral bleeding; leucocytes; autoaggressive T-cells; acute media infarct or acute intracerebral bleeding
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples (serum and plasma)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with acute media infarct
- controls with cardiovascular risks

SUMMARY:
The damage of the brain parenchyma, as well as the stroke-induced dysfunction of the blood-brain-barrier can make previously hidden CNS antigens "visible", and can thus lead to the development of autoimmune mechanisms.

It seems plausible that stroke-associated immunodepression influences the development and the phenotype of these autoreactive immune responses.

This study will investigate whether cerebral ischemia leads to changes in the immune response, in particular to the development and/or proliferation of autoreactive effector T-cells and/or regulatory T-cells. Furthermore, the association between the severity and the phenotype of this autoimmune response and the clinical course, i.e. prognosis and mortality, will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* acute media infarct or intracerebral bleeding within the last 36 h (patients)
* NIHSS > 7 (patients)
* age > 17 years (patients), age > 54 years (controls)
* informed consent of patient or legal representative/ of control
* cardiovascular risk such as diabetes mellitus (control)

Exclusion Criteria:

* infections (patients, controls)
* antibiotic or immunosuppressive treatment within the last 4 weeks (patients)
* other CNS disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: acute media infarct or intracerebral bleeding
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2009-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
autoantigen-specific T-cells in patients with acute media infarct | within 36 h
  quantitative determination of autoantigen-specific T-cells in patients with acute media infarct
leukocytes in patients with acute media infarct | within 36 hours
  quantitative and qualitative analysis of leukocytes in patients with acute media infarct

SECONDARY OUTCOMES:
frequency and phenotype of CNS-autoreactive immune cells under the influence of immunodepression | within 36 h, after day 3, 7, 90 and 180
clinical course, i.e. mortality and prognosis (measured by mod. Rankin Scale) | after day 90 and 180
clinical course, i.e. mortality and prognosis (measured by Bartel Index) | after day 90 and 180

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meisel, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Result] Klehmet J, Hoffmann S, Walter G, Meisel C, Meisel A. Stroke induces specific alteration of T memory compartment controlling auto-reactive CNS antigen-specific T cell responses. J Neurol Sci. 2016 Sep 15;368:77-83. doi: 10.1016/j.jns.2016.06.039. Epub 2016 Jun 17. PMID 27538605